CLINICAL TRIAL: NCT02323620
Title: The Impact of Repeated Intracoronary Injection of Autologous Bone-marrow Derived Mononuclear Cells for Left Ventricle Contractility and Remodeling in Patients With STEMI.Prospective Randomized Study.
Brief Title: Impact of Intracoronary Injection of Autologous BMMC for LV Contractility and Remodeling in Patients With STEMI
Acronym: RACE-STEMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Heart of Poland (Other)
Responsible Party: Principal Investigator, Pawel Buszman, MD, PhD, American Heart of Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHP-001
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2018-12

CONDITIONS: Heart Failure; Myocardial Infarction
Keywords: Acute myocardial Infarction; bone marrow; stem cells; cardiovascular disease; mortality
MeSH Terms: conditions — Heart Failure; Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Optimal standard care after myocardial infarction.
- Intracoronary infusion of BM-MC (Experimental): Bone marrow-derived progenitor autologous cells aspiration and intracoronary infusion of the cells.
  Interventions: Procedure: Intracoronary infusion of BM-MC

INTERVENTIONS:
Procedure: Intracoronary infusion of BM-MC — Bone marrow-derived progenitor cells are obtained from 60ml bone marrow aspirated from the iliac crest. Intracoronary infusion of the autologous cells is performed via conventional percutaneous intracoronary intervention techniques using an over-the-wire balloon technique.
  Arms: Intracoronary infusion of BM-MC

SUMMARY:
This is multicentre, randomised open-label, controlled, parallel-group phase III study. Its aim is to demonstrate that a triple intracoronary infusion of autologous bone marrow-derived mononuclear cells in addition to state of the art treatment is safe and reduces all-cause mortality in patients with reduced left ventricular ejection fraction (≤45%) after successful reperfusion for acute myocardial infarction when compared to a control group of patients undergoing best medical care.

DETAILED DESCRIPTION:
The study is divided into 3 parts:

* Screening phase: Patients will be recruited at the investigational clinical centers. Alternatively, patients who had primary PCI performed at institutions different from the investigational sites can also be enrolled. Interested patients may be referred for screening to any of the participating study sites after acute reperfusion therapy. Informed consent and assessment of eligibility of patients with respect to in- and exclusion criteria will be done at the investigational site. If all other eligibility criteria are met, echocardiography will be performed 3 to 6 days after the acute PCI, and ejection fraction will be quantified by a central Echo Core Lab after web based transmission. CT examination will be performed 1 month after acute PCI in all screened patients with LVEF ≤ 45%. If LVEF will not improve ≥5% in the CT the patient may be qualified into the Study.
* Treatment phase: Bone marrow aspiration will be performed for the patients assigned to the treatment group (II). Bone marrow will be collected from the patient and MNC isolated using point-of-care system (Harvest) at a Site. Intracoronary infusion of BM-MNCs will be performed up to 2 hours after isolation via radial approach. Same procedure will be performed 3 and 6 months after first application.
* Follow-up phase: After hospital discharge, patients will be followed up per telephone 30 days and 3, 6, 9 months after randomisation and with a site visit with CT examination 12 months after randomisation. Afterwards, telephone follow up will be performed every 3 months. Once the required number of clinical events has been observed, all patients will attend a final study visit, but minimum follow up period for each patient is 2 years. Endpoints will be reported as occurring throughout the follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women of any ethnic origin aged ≥ 18 years.
2. Patients with acute ST-elevation myocardial infarction as defined by the universal definition of AMI.
3. Successful acute reperfusion therapy (residual stenosis visually <50% and TIMI flow ≥2) within 24 hours of symptom onset or thrombolysis within 12 hours of symptom onset followed by successful percutaneous coronary intervention (PCI) within 24 hours after thrombolysis.
4. Left ventricular ejection fraction ≤ 45% with significant regional wall motion abnormality assessed by quantitative echocardiography (central, independent core lab analysis) 3 to 6 days after reperfusion therapy
5. Open coronary artery suitable for cell infusion supplying the target area of abnormal wall motion
6. LVEF≤45% with significant regional wall motion abnormality assessed by computed tomography (CT) 30 days after reperfusion therapy with no LVEF improvement ≥5%.

Exclusion Criteria:

1. Participation in another clinical trial within 30 days prior to randomisation
2. Previously received stem/progenitor cell therapy
3. Pregnant or nursing women
4. Mental condition rendering the patient unable to understand the nature, scope and possible consequences of the study or to follow the protocol
5. Necessity to revascularise additional vessels, outside the target coronary artery at the time of BM-MNC infusion (additional revascularisations after primary PCI and before BM-MNC cell infusion are allowed)
6. Cardiogenic shock requiring mechanical support
7. Platelet count <100,000/μl, or hemoglobin <8.5 g/dl
8. Impaired renal function, i.e. serum creatinine >2.5 mg/dl
9. Persistent fever or diarrhea not responsive to treatment within 4 weeks prior screening
10. Clinically significant bleeding within 3 months prior screening
11. Uncontrolled hypertension (systolic >180 mmHg and diastolic >120 mmHg)
12. Life expectancy of less than 2 years from any non-cardiac cause or neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricle ejection fraction change evaluated by CT | 12 months

SECONDARY OUTCOMES:
Change in left ventricle End-Systolic Volume (ESV) and End-Diastolic Volume (EDV) evaluated by CT | 12 months
Time from randomisation to cardiac death | 3 years
Time from randomisation to cardiovascular death or rehospitalisation due to heart failure | 3 years
Incidence and severity of adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pawel E Buszman, MD, PhD, Principal Investigator — American Heart of Poland
Locations (1):
- Polsko-Amerykańskie Kliniki Serca, Ustroń, Poland